CLINICAL TRIAL: NCT05020886
Title: Evaluation and Improving Strategy of Turning Performance in Individuals With Stroke
Brief Title: Turning Performance in Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Other Study IDs: YM109175E
Record Dates: First submitted 2021-08-21; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy
  Interventions: Behavioral: turning task
- Stroke
  Interventions: Behavioral: turning task

INTERVENTIONS:
Behavioral: turning task — Several trials included bilateral turning in 30, 60, 90, 120, 150, 180 degree.

SUMMARY:
Turning is a challenging task for stroke patient. Previous studies showed that turning is one of the activities which resulting in falling frequently in stroke. However, the assessment tool of turning performance is still lack of reliability and validity. Furthermore, the main factors which affected turning ability in stroke are not approved yet.

ELIGIBILITY:
Inclusion Criteria:

* 6 months after first stroke.
* Able to independently walk 7 meter at least without any device
* MMSE score ≧ 24

Exclusion Criteria:

* Unstable medical conditions (such as deep vein thrombosis)
* Any disease which has known affecting walk(heart failure, diabetes)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Turning angle | 10 minutes
Turning time | 10 minutes
Turning step | 10 minutes
Single leg supported time during turning | 10 minutes
Swing time during turning | 10 minutes